CLINICAL TRIAL: NCT04351178
Title: F@ce 2.0 - Implementation and Evaluation of a Model for a Person-centred, Information and Communication Technology and Team Based Rehabilitation Intervention for People Who Have Had Stroke in Sweden
Brief Title: F@ce 2.0 - Information and Communication Technology-based Rehabilitation Intervention After Stroke in Sweden
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Forte (Industry)
Responsible Party: Principal Investigator, Susanne Guidetti, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HELD, Karolinska Institutet
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to participate in F@ce 2.0 (IG) or a control group (CG) receiving usual rehabilitation at two different sites; both an urban (IG+CG) and rural site (CG+IG) in Sweden
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile phone supported and team based rehabilitation (Experimental): Participants in the intervention group will receive an 8-week mobile phone supported and team based rehabilitation intervention (F@ce 2.0)
  Interventions: Behavioral: Mobile phone supported and team based rehabilitation
- Rehabilitation as usual (Active Comparator): Control group participants will receive rehabilitation as usual and in addition information about stroke.
  Interventions: Behavioral: Rehabilitation as usual

INTERVENTIONS:
Behavioral: Mobile phone supported and team based rehabilitation — Participants in the intervention group will receive an 8-week mobile phone supported and team based rehabilitation intervention (F@ce 2.0).The participants will be introduced to a problem-solving strategy intended to facilitate the learning and problem-solving process to be used during the intervention. The strategy will provide a structure for healthcare professionals delivering the intervention. Three goals in daily activities will be formulated that the person wants and needs to do within the home environment. Each activity will be practiced together with the healthcare professionals and significant others. The significant others will be informed about the participant's goals and the planned strategies for reaching the goals. The participants will practice the activities in their home environment supported by mobile phone calls and text messages. In addition they will be given information about stroke.
  Arms: Mobile phone supported and team based rehabilitation
Behavioral: Rehabilitation as usual — Control group participants will receive rehabilitation as usual and in addition information about stroke.
  Arms: Rehabilitation as usual

SUMMARY:
The purpose of the present proposal is to implement and evaluate a new model for mobile phone supported and family-centred rehabilitation intervention (F@ce 2.0) with regard to functioning in activities in daily living and participation in everyday life among persons with stroke and their families in rural and urban areas in Sweden.

DETAILED DESCRIPTION:
The investigators' previous feasibility study suggested beneficial effects on occupational performance and satisfaction of a mobile phone supported and person-centred rehabilitation intervention (F@ce1.0) after stroke in Stockholm, Sweden. The purpose of the present proposal is to implement and evaluate F@ce 2.0 on functioning in activities in daily living (ADL) and participation in everyday life among persons with stroke and their significant others (someone identified by the person with stroke as close i.e.partner, friend, son, daughter).

With recommendations on evaluation of complex interventions both outcomes and processes will be studied and hence both quantitative and qualitative methods will be applied. In a randomized controlled trial F@ce 2.0 will be evaluated compared to ordinary rehabilitation in urban/rural Sweden regarding; self-efficacy, perceived performance and participation in everyday activities, independence in ADL, health care utilization and the families´ perceived participation in everyday activities. Qualitative data will explore experiences of people with stroke, significant others and rehabilitation staff of participating in F@ce 2.0. The research project has a multidisciplinary perspective for sustainable rehabilitation interventions, a prerequisite for better participation in everyday life for people with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have had a stroke
* Enrolled in one of the participating home rehabilitation teams in Stockholm and Dalarna
* Able to participate in eight weeks of intervention

Exclusion Criteria:

* Inability to formulate activity goals
* Inability to express themselves in Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Self-efficacy Scale | Change between enrollment, after the 8 weeks of intervention and 6 months after enrollment
  Participants are instructed to rate how confident they feel about performing each of 16 everyday activities on a 10-point rating scale ranging from 1) "not confident at all in my ability" to 10) "very confident in my ability". The average of all responses are calculated
Canadian Occupational Performance Measure (COPM) | Change between enrollment, after the 8 weeks of intervention and 6 months after enrollment
  Canadian Occupational Performance Measure (COPM) measures performance and satisfaction in self-care, productivity and leisure from the individual's perspective. The participant is asked 1) to rate performance of the specified activities using a 1 (low) to 10 (high) scale and 2) to score his or her satisfaction with that performance using the same scale. Weighted scores of the chosen activities are added separately for performance and satisfaction to create two summative scores. The summative scores are then divided by the number of rated activities to provide COPM scores.
Caregiver Burden Scale | Change between enrollment, after the 8 weeks of intervention and 6 months after enrollment
  Questionnaire that consists of 22 items for different types of subjective caregiver burden, covering areas of the caregiver's health, feelings of psychological well-being, relations, social network, physical workload, and environmental aspects. The items are scored on a scale from 1 to 4 and the higher the score the greater the burden.

SECONDARY OUTCOMES:
Stroke Impact Scale (SIS) 3.0 | Change between enrollment, after the 8 weeks of intervention and 6 months after enrollment
  Assesses the perceived impact on functioning in everyday life in eight domains: Strength, Memory and thinking, Emotions, Communication, ADL/ Instrumental activities of daily living (IADL), Mobility, Hand function and Participation. The SIS includes 59 items within these eight domains. Aggregated scores ranges from 0 to 100, the higher the score, the lower the perceived impact of stroke, i.e. fewer problems in everyday life. The SIS 3.0 also includes a question to assess the participant's global perception of recovery presented in a vertical analogue scale ranging from '0 = no recovery to 100 = full recovery'
Frenchay Activities Index | Change between enrollment, after the 8 weeks of intervention and 6 months after enrollment
  Questionnaire consisting of 15 items on frequency of social everyday activities and the score is based on the frequency with which an activity has been performed during the previous 3 or 6 months. The total score ranges from 0 (inactive) to 45 (very active).
Fatigue Severity Scale-7 | Change between enrollment, after the 8 weeks of intervention and 6 months after enrollment
  Questionnaire that assesses fatigue. The final score is the mean of the seven items graded between 1 (strongly disagree) and 7 (strongly agree). Scores are categorized as no fatigue (1-3) or fatigue (4-7)
Hospital Anxiety and Depression Scale | Change between enrollment, after the 8 weeks of intervention and 6 months after enrollment
  Questionnaire that assesses anxiety and depression comprising two subscales, each ranging from 0-21. Scores are categorised as no anxiety and depression (0-7), mild (8-10) or moderate to severe anxiety and depression (10-21)
Life Satisfaction Checklist | Change between enrollment, after the 8 weeks of intervention and 6 months after enrollment
  Questionnaire that assesses life satisfaction with the global item "Life as a whole" and ten domain specific items. Answering alternatives range from 1 (very dissatisfied) to 6 (very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Guidetti, Professor, Principal Investigator — Karolinska Institutet
Locations (12):
- Sweden (12):
  - Primärvårdsrehab Bromma, Stockholms Sjukhem, Stockholm, Bromma
  - Neuroteam Värmdö Rehab, Stockholm, Gustavsberg
  - Aleris Rudans rehab Haninge, Stockholm, Handen
  - Aleris Rehab Skärholmen Neuroteam, Stockholm, Skärholmen
  - Avesta, Avesta
  - Borlänge hemrehab, Borlänge
  - Falun hemrehab, Falun
  - Externa stroketeamet Gävle, Gävle
  - Externa stroketeamet Hudiksvall, Hudiksvall
  - Mora hemrehab, Mora
  - Neuroteam Kungsholmen, Stockholms sjukhem, Stockholm
  - Aleris Rehab Älvsjö Neuroteam, Stockholm, Älvsjö

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soderhielm K, Tistad M, Ytterberg C, Guidetti S. Experiences of F@ce 2.0: a person-centred intervention for home-based rehabilitation after stroke supported by digital technology - a qualitative study. BMJ Open. 2025 Jul 16;15(7):e089147. doi: 10.1136/bmjopen-2024-089147. PMID 40669890
- [Derived] Eriksson G, Tistad M, Elf M, Fors U, von Koch L, Ytterberg C, Guidetti S. Study protocol of a non-randomised controlled trial evaluating the effectiveness of the F@ce 2.0 programme: a person-centred, ICT-supported and interdisciplinary rehabilitation intervention after stroke. BMJ Open. 2022 Aug 4;12(8):e058748. doi: 10.1136/bmjopen-2021-058748. PMID 35926996